CLINICAL TRIAL: NCT02921100
Title: A Prospective Comparison of Digital Image Analysis and Routine Cytology for the Identification of Pancreatic Neoplasia in Patient Undergoing EUS-FNA
Brief Title: Comparison of DNA Ploidy and Conventional Cytology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of gastroenterology department, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DNA ploidy and CC
Record Dates: First submitted 2016-09-26; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Biopsy, Fine-Needle
MeSH Terms: interventions — Cytological Techniques; Ploidies; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional cytology (Other): Patients in this arm will undergo an operation of EUS-FNA . The acquired cytological samples from EUS-FNA will undergo a conventional cytology.
  Interventions: Procedure: cytology; Procedure: EUS-FNA; Device: EUS-guided fine needle
- DNA ploidy test (Other): Patients in this arm will undergo an operation of EUS-FNA . The acquired cytological samples from EUS-FNA will undergo DNA ploidy test.
  Interventions: Procedure: DNA ploidy; Procedure: EUS-FNA; Device: EUS-guided fine needle

INTERVENTIONS:
Procedure: cytology — The conventional cytology was interpreted independently by two cytopathologists, both of whom are blinded to the DIA results. The conventional cytologic diagnosis were classified as no abnormal cells, atypical cells, suspicious malignant cells and malignant cells.
  Arms: Conventional cytology
Procedure: DNA ploidy — DIA is a form of cytologic analysis that quantifies cellular constituents by using spectro photometric principles and a sister technique to flow cytometry.Quantification of DNA content, chromatin distribution, and nuclear morphology can be determined and suggest features of malignancy
  Other Names: digital image analysis
  Arms: DNA ploidy test
Procedure: EUS-FNA — All the enrolled participants underwent an operation of EUS-guided fine needle aspiration. Histological and cytological samples were obtained following this step.
Device: EUS-guided fine needle

SUMMARY:
150 patients who had suspected pancreatic malignancy were planed to be enrolled in this study. Equal cytological samples of each patient undergoing EUS-FNA were examined by digital image analysis and conventional cytology respectively. The investigators aim to compare the efficacy of DIA and conventional cytology in diagnosing pancreatic cancer. Further more, the investigators also collected the blood sample of each enrolled patient for advanced study.

DETAILED DESCRIPTION:
The conventional cytology was interpreted independently by two cytopathologists, both of whom are blinded to the DIA results. The conventional cytologic diagnosis were classified as no abnormal cells, atypical cells, suspicious malignant cells and malignant cells. The specimens were examined by two experienced cytopathologists. Any disagreement on specimens would refer to a third cytopathologist to provide a final consensus. The former two diagnosis were determined to be positive, and the latter two to be negative.

DIA is a form of cytologic analysis that quantifies cellular constituents by using spectro photometric principles and a sister technique to flow cytometry. Computer analysis of the pixels produces a digital image of the nucleus and other cellular constituents. Quantification of DNA content, chromatin distribution, and nuclear morphology can be determined and suggest features of malignancy. ThinPrep specimens were prepared as previously described.Per specimen, the DNA content of at least 500 cells was selected for quantification using an image analyzer (Landing Medical High-tech, Wuhan, Hubei, China) and the mean integrated optical density lymphocytes served as an internal standard control. All other histograms suggesting the presence of (1) any cells with DNA>5c; (2) diploidy cells with a very high proliferation rate where 10% or more of the total cells were found in the proliferation fraction; and (3) a population of aneuploidy stem cells, were called positive for malignancy. Images of cells reporting a DNA amount greater than 5c were examined microscopically by a cytotechnologist to exclude any artifacts such as dust, air bubbles, overlapping cells, etc. from the >5c cell galleries.

All the final diagnosis are to be confirmed by histopathology or a long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. who had known or suspected pancreatic malignancy and
2. in whom the endosonographer deemed the target lesion safe and feasible to allow the necessary study passes.

Exclusion Criteria:

1. not willing to sign informed consent,
2. cells obtained from FNA for DNA ploidy test less than 200, and/or
3. patients do not cooperate with follow-up.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with accurate diagnosis by conventional cytology versus by DNA ploidy test | 12 months

SECONDARY OUTCOMES:
sensitivity of conventional cytology Versus DNA ploidy test in the diagnosis of pancreatic malignancy | 12 months
specificity of conventional cytology Versus DNA ploidy test in the diagnosis of pancreatic malignancy | 12 months
positive predictive value of conventional cytology Versus DNA ploidy test in the diagnosis of pancreatic malignancy | 12 months
negative predictive value of conventional cytology Versus DNA ploidy test in the diagnosis of pancreatic malignancy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wang, Dr., Study Director — Digestive endoscopic center of Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No